CLINICAL TRIAL: NCT01505556
Title: Proprioceptive Postural Control and Diaphragm Paresis
Status: Withdrawn | Type: Observational
Why Stopped: Problems to recruit individuals with diaphragm paresis.
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Simon Brumagne, Prof. dr. Simon Brumagne, KU Leuven
Other Study IDs: 2012_SBrumagne_DiaphParesis; 1.5.104.03, G.0674.09 (Other Grant/Funding Number: Research Foundation Flanders (FWO))
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Proprioceptive Postural Control; Respiratory Disorders; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Respiration Disorders; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Diaphragm paresis
- Healthy controls

SUMMARY:
Proprioceptive weighting changes may explain differences in postural control performance. In addition, the respiratory movement has a disturbing effect on postural balance. Postural balance seems to be impaired in individuals with respiratory disorders. Increased risk of falling is reported in individuals with chronic obstructive pulmonary disease. Besides the essential role of respiration, the diaphragm may also play an important role in the control of the trunk and postural balance.

The aim of the study is to clarify whether proprioceptive postural control is impaired in individuals with diaphragm paresis.

ELIGIBILITY:
Inclusion Criteria individuals with diaphragm paresis:

* Age: 18-70 years old
* Unilateral or bilateral diaphragm paresis following paresis of phrenic nerve
* Willingness to sign the informed consent

Inclusion Criteria healthy controls:

* Age: 18-70 years old
* Spirometry: FEV1/FVC ≥ 0.7 and FEV1 > 80%
* Willingness to sign the informed consent

Exclusion Criteria:

* History of major trauma and/or major orthopedic surgery of the spine, the pelvis or the lower quadrant
* One of the following conditions: Parkinson, multiple sclerosis, stroke, history of vestibular disorder
* Respiratory disorder other than diaphragm paresis
* Recent diagnosis of cancer
* Significant cardiovascular comorbidity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients from the University Hospital Leuven - Respiratory Disvision
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Proprioceptive postural control | 1 year
  Center of pressure displacement (force plate) in standing in response to local muscle vibration on ankle and back muscles to specifically detect the role of proprioception in postural control.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Brumagne, PhD, Principal Investigator — KU Leuven; Thierry Troosters, PhD, Principal Investigator — KU Leuven; Wim Janssens, MD, PhD, Principal Investigator — KU Leuven; Marc Decramer, MD, PhD, Principal Investigator — KU Leuven
Locations (1):
- Katholieke Universiteit Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Background] Janssens L, Brumagne S, Polspoel K, Troosters T, McConnell A. The effect of inspiratory muscles fatigue on postural control in people with and without recurrent low back pain. Spine (Phila Pa 1976). 2010 May 1;35(10):1088-94. doi: 10.1097/BRS.0b013e3181bee5c3. PMID 20393397